CLINICAL TRIAL: NCT00650468
Title: A Prospective, Randomized, Multi-Center Double-Blind Study of Early Corticosteroid Cessation vs. Long Term Corticosteroid Therapy With Prograf and CellCept in Primary Renal Transplant Patients
Brief Title: A Study to Compare Early Steroid Withdrawal and Long-Term Steroid Maintenance Therapy in Kidney Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sr. Manager Clinical Trail Registry, Astellas Pharma US, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-99-001
Record Dates: First submitted 2008-03-17; First posted 2008-04-01 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2009-03

CONDITIONS: Renal Transplantation
Keywords: Renal Transplantation; Prograf
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid; Steroids; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): early steroid cessation
  Interventions: Drug: tacrolimus; Drug: CellCept; Drug: steroids (methylprednisone or prednisone)
- 2 (Experimental): long-term maintenance steroids
  Interventions: Drug: tacrolimus; Drug: CellCept; Drug: steroids (methylprednisone or prednisone)

INTERVENTIONS:
Drug: tacrolimus — Oral
  Other Names: Prograf; FK506
Drug: CellCept — IV or Oral
  Other Names: MMF; Mycophenolate mofetil
Drug: steroids (methylprednisone or prednisone) — IV or Oral
  Other Names: methylprednisone; prednisone

SUMMARY:
A study comparing the early withdrawal of steroids to long-term maintenance steroid therapy in Kidney Transplant Patients receiving Prograf and Cellcept

ELIGIBILITY:
Inclusion:

* Patient is between post kidney transplant day 3-7 and no requirement for dialysis

Exclusion:

* Patient is receiving kidney from HLA identical,living donor
* Patient is a multi-organ transplant recipient
* Patient is pregnant or lactating. Female patients of child bering potential must have a negative pregnancy test and agree to practice effective birth control

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 1999-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Assessment of death, graft loss, or severe acute rejection | 6 months, 12 months, yearly up to 5 years

SECONDARY OUTCOMES:
Comparison of patient and graf survival | 6 months, 12 months, yearly up to 5 years
Incidence and severity of acute rejection | 6 months, 12 months, yearly up to 5 years
Need for antilymphocyte treatment | 6 months, 12 months, yearly up to 5 years
Graft function | 6 month, 12 months, yearly up to 5 years
Framingham Coronary Heart Disease Risk Factors | 6 months, 12 months, yearly up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: central contact, Study Director — Astellas Pharma US, Inc.
Locations (27):
- United States (27):
  - Little Rock, Arkansas
  - Loma Linda, California
  - Los Angeles, California
  - Denver, Colorado
  - Chicago, Illinois
  - Lexington, Kentucky
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - Omaha, Nebraska
  - New Brunswick, New Jersey
  - Buffalo, New York
  - New York, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Providence, Rhode Island
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Galveston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Madison, Wisconsin
  - Milwaukee, Wisconsin

REFERENCES:
- [Background] Woodle ES; Fujisawa Corticosteroid Withdrawal Study Group. A prospective, randomized, multicenter, double-blind study of early corticosteroid cessation versus long-term maintenance of corticosteroid therapy with tacrolimus and mycophenolate mofetil in primary renal transplant recipients: one year report. Transplant Proc. 2005 Mar;37(2):804-8. doi: 10.1016/j.transproceed.2004.12.083. PMID 15848538
- [Background] Woodle ES, First MR, Pirsch J, Shihab F, Gaber AO, Van Veldhuisen P; Astellas Corticosteroid Withdrawal Study Group. A prospective, randomized, double-blind, placebo-controlled multicenter trial comparing early (7 day) corticosteroid cessation versus long-term, low-dose corticosteroid therapy. Ann Surg. 2008 Oct;248(4):564-77. doi: 10.1097/SLA.0b013e318187d1da. PMID 18936569
- [Derived] Gaber AO, Moore LW, Alloway RR, Woodle ES, Pirsch J, Shihab F, Henning A, Fitzsimmons W, Holman J, Reisfield R, First MR; Astellas Corticosteroid Withdrawal Study Group. Acute rejection characteristics from a prospective, randomized, double-blind, placebo-controlled multicenter trial of early corticosteroid withdrawal. Transplantation. 2013 Feb 27;95(4):573-9. doi: 10.1097/TP.0b013e3182777efb. PMID 23423269
- [Derived] Delgado JC, Fuller A, Ozawa M, Smith L, Terasaki PI, Shihab FS, Eckels DD. No occurrence of de novo HLA antibodies in patients with early corticosteroid withdrawal in a 5-year prospective randomized study. Transplantation. 2009 Feb 27;87(4):546-8. doi: 10.1097/TP.0b013e3181949d2e. PMID 19307792